CLINICAL TRIAL: NCT03323346
Title: Phase II Open Labeled Trial of Disulfiram With Copper in Metastatic Breast Cancer
Brief Title: Phase II Trial of Disulfiram With Copper in Metastatic Breast Cancer
Acronym: DISC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1-DSF-MBC
Record Dates: First submitted 2017-09-29; First posted 2017-10-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasm Female; Metastatic Breast Cancer
Keywords: metastatic breast cancer; disulfiram; cooper
MeSH Terms: conditions — Breast Neoplasms | interventions — Disulfiram; Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disulfiram with copper (Experimental): Patients will take one pill of disulfiram (Antabus) daily at a dose of 400 mg continually during the treatment phase (from day 0 till End of treatment Visit). In case of intolerance, lower dose up to 200 mg per day is allowed. Patients will take disulfiram after their evening meal.
  Patients will avoid alcohol and other disulfiram-drug interactions will be considered.
  Copper supplementation will be given separately from disulfiram; in the morning with patients´breakfast. Patients will take one pill of copper dietary supplement (for instance Copper Star, STARLIFE) corresponding to 2 mg of elementary copper.
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Patients will take one pill of disulfiram (Antabus) daily at a dose of 400 mg continually during the treatment phase (from day 0 till End of treatment Visit). In case of intolerance, lower dose up to 200 mg per day is allowed.
  Copper supplementation will be given separately from disulfiram; in the morning with patients´breakfast. Patients will take one pill of copper dietary supplement (for instance Copper Star, STARLIFE) corresponding to 2 mg of elementary copper.
  Other Names: Copper

SUMMARY:
The aim of the study is to establish clinical evidence for introducing disulfiram and cooper as an active therapy for metastatic breast cancer upon failure of conventional systemic and/or locoregional therapies.

Analyses of the following objectives will be performed in the population of patients with metastatic breast cancer:

Primary efficacy objective:

To evaluate the efficacy of the treatment by assessment of:

* clinical response rate (RR)
* clinical benefit rate (CBR)

Secondary efficacy objectives:

To evaluate the efficacy of the treatment by assessment of:

* time to progression (TTP)
* overall survival (OS)

Pharmacokinetic objectives:

• to determine pharmacokinetic parameters for disulfiram and its active metabolites administered in combination with copper supplements in cancer patient population

Safety objectives:

• to describe safety profile of disulfiram administered in combination with copper supplements

Exploratory objectives:

Parallel analysis to assess (identify) potential candidate surrogate biomarkers of disulfiram efficacy, as well as identification (using proteomic, biochemical and molecular genetic studies) of potential predictive biomarkers of disulfiram sensitivity or resistance will be performed. Surrogate biomarker analysis will focus on in vivo ubiquitin-proteosomal system inhibition, cell cycle and DNA damage.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Patients with stage IV breast cancer with metastases demonstrated by appropriate imaging techniques
2. Histologically or cytologically confirmed tumor
3. Age of 18 years or more
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
5. Patients have failed, untolerated or refused standard therapeutic modalities
6. Not received systemic anticancer therapy or radiation or had major surgery in last 2 weeks
7. Not currently participating in another study
8. Anticipated survival of at least 2 months
9. Baseline aspartate aminotransferase (AST) and alanine aminotransferase (ALT) not greater than 2.5 X upper institutional limit
10. Serum copper within normal limits
11. Serum ceruloplasmin > 17 mg/dL
12. Able and willing to sign informed consent and to comply with study procedures
13. Able to ingest oral medications
14. No known allergy to disulfiram or copper
15. Willing to refrain from ingestion of alcoholic beverages while on the study

Exclusion criteria:

1. Participation in another clinical trial of a therapeutic drug during the past 14 days
2. Addiction to alcohol or drugs
3. Baseline AST or ALT greater than 2.5 X upper institutional limit
4. Unable to ingest oral medications
5. Unable to undergo CT/SPECT scanning because of inability to lie recumbent in the scanner
6. Actively receiving cytotoxic cancer chemotherapy agents
7. Anticipated survival of less than 2 months
8. Women of child-bearing potential who are not using a commonly accepted effective means of contraception; women of child-bearing potential will have negative pregnancy test before enrollment
9. History of active liver disease, including chronic active hepatitis, viral hepatitis (hepatitis B, C and CMV), cholestatic jaundice of any etiology, toxic hepatitis, or cholestatic hepatitis or jaundice with bilirubin greater than 2.0 X upper institutional limit
10. History of Wilson's disease or family member with Wilson's disease
11. History of hemochromatosis or family member with hemochromatosis
12. History of other iron overload syndrome such as hemochromatosis
13. Need for metronidazole, warfarin and/or theophylline medication, the metabolism of which is likely influenced by disulfiram
14. Pregnant women and nursing mothers are not allowed to enroll on this study
15. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IV breast cancer with metastases demonstrated by appropriate imaging techniques (computer tomography - CT, positron emission tomography - PET or PET/CT, MRI, ultrasound, etc.)
2. Histologically or cytologically confirmed tumor
3. Age of 18 years or more
4. ECOG performance status of 0 - 2
5. Patients have failed, untolerated or refused standard therapeutic modalities
6. Not received systemic anticancer therapy or radiation or had major surgery in last 2 weeks
7. Not currently participating in another study
8. Anticipated survival of at least 2 months
9. Baseline AST and ALT not greater than 2.5 X upper institutional limit
10. Serum copper within normal limits
11. Serum ceruloplasmin > 17 mg/dL
12. Able and willing to sign informed consent and to comply with study procedures
13. Able to ingest oral medications
14. No known allergy to disulfiram or copper
15. Willing to refrain from ingestion of alcoholic beverages while on the study

Exclusion Criteria:

1. Participation in another clinical trial of a therapeutic drug during the past 14 days
2. Addiction to alcohol or drugs
3. Baseline AST or ALT greater than 2.5 X upper institutional limit
4. Unable to ingest oral medications
5. Unable to undergo CT/SPECT scanning because of inability to lie recumbent in the scanner
6. Actively receiving cytotoxic cancer chemotherapy agents
7. Anticipated survival of less than 2 months
8. Women of child-bearing potential who are not using a commonly accepted effective means of contraception; women of child-bearing potential will have negative pregnancy test before enrollment
9. History of active liver disease, including chronic active hepatitis, viral hepatitis (hepatitis B, C and CMV), cholestatic jaundice of any etiology, toxic hepatitis, or cholestatic hepatitis or jaundice with bilirubin greater than 2.0 X upper institutional limit
10. History of Wilson's disease or family member with Wilson's disease
11. History of hemochromatosis or family member with hemochromatosis
12. History of other iron overload syndrome such as hemochromatosis
13. Need for metronidazole, warfarin and/or theophylline medication, the metabolism of which is likely influenced by disulfiram
14. Pregnant women and nursing mothers are not allowed to enroll on this study
15. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate (RR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  sum of complete and partial responses (CR+PR)
Clinical benefit rate (CBR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  sum of complete, partial responses and stable diseases (CR+PR)CR+PR+SD)

SECONDARY OUTCOMES:
Time to progression (TTP) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  time to progression (TTP) in months
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  overall survival (OS) in months
The pharmacokinetic (PK) characteristics | Day 0 = at first administration of the drug
  Cmax
The pharmacokinetic (PK) characteristic - Area Under Curve (AUC) | Day 0 = at first administration of the drug
  AUC - The area under the plasma concentration over the time
The pharmacokinetic (PK) characteristic - T-max | Day 0 = at first administration of the drug
  T-max - Time to reach maximum concentration
The pharmacokinetic (PK) characteristic - T1/2 | Day 0 = at first administration of the drug
  T1/2 - Apparent terminal elimination half-life time
The pharmacokinetic (PK) characteristic - λz | Day 0 = at first administration of the drug
  λz (Lambda-z) - Individual estimate of the terminal elimination rate constant, calculated using log-linear regression of the terminal portions of the plasma concentration-versus-time curves
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of participants with treatment-related adverse events analyzed as cumulative burden at every 6 months until study termination.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD., PhD., Study Chair — Palacky University
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Askgaard G, Friis S, Hallas J, Thygesen LC, Pottegard A. Use of disulfiram and risk of cancer: a population-based case-control study. Eur J Cancer Prev. 2014 May;23(3):225-32. doi: 10.1097/CEJ.0b013e3283647466. PMID 23863824
- [Background] Wickstrom M, Danielsson K, Rickardson L, Gullbo J, Nygren P, Isaksson A, Larsson R, Lovborg H. Pharmacological profiling of disulfiram using human tumor cell lines and human tumor cells from patients. Biochem Pharmacol. 2007 Jan 1;73(1):25-33. doi: 10.1016/j.bcp.2006.08.016. Epub 2006 Aug 26. PMID 17026967
- [Background] Schweizer MT, Lin J, Blackford A, Bardia A, King S, Armstrong AJ, Rudek MA, Yegnasubramanian S, Carducci MA. Pharmacodynamic study of disulfiram in men with non-metastatic recurrent prostate cancer. Prostate Cancer Prostatic Dis. 2013 Dec;16(4):357-61. doi: 10.1038/pcan.2013.28. Epub 2013 Aug 20. PMID 23958896
- [Background] Brar SS, Grigg C, Wilson KS, Holder WD Jr, Dreau D, Austin C, Foster M, Ghio AJ, Whorton AR, Stowell GW, Whittall LB, Whittle RR, White DP, Kennedy TP. Disulfiram inhibits activating transcription factor/cyclic AMP-responsive element binding protein and human melanoma growth in a metal-dependent manner in vitro, in mice and in a patient with metastatic disease. Mol Cancer Ther. 2004 Sep;3(9):1049-60. PMID 15367699
- [Background] Lewison EF. Spontaneous regression of breast cancer. Prog Clin Biol Res. 1977;12:47-53. No abstract available. PMID 918117
- [Background] Lin J, Haffner MC, Zhang Y, Lee BH, Brennen WN, Britton J, Kachhap SK, Shim JS, Liu JO, Nelson WG, Yegnasubramanian S, Carducci MA. Disulfiram is a DNA demethylating agent and inhibits prostate cancer cell growth. Prostate. 2011 Mar 1;71(4):333-43. doi: 10.1002/pros.21247. Epub 2010 Aug 31. PMID 20809552
- [Background] Robinson TJ, Pai M, Liu JC, Vizeacoumar F, Sun T, Egan SE, Datti A, Huang J, Zacksenhaus E. High-throughput screen identifies disulfiram as a potential therapeutic for triple-negative breast cancer cells: interaction with IQ motif-containing factors. Cell Cycle. 2013 Sep 15;12(18):3013-24. doi: 10.4161/cc.26063. Epub 2013 Aug 12. PMID 23974104
- [Background] Cvek B, Milacic V, Taraba J, Dou QP. Ni(II), Cu(II), and Zn(II) diethyldithiocarbamate complexes show various activities against the proteasome in breast cancer cells. J Med Chem. 2008 Oct 23;51(20):6256-8. doi: 10.1021/jm8007807. Epub 2008 Sep 25. PMID 18816109
- [Background] Chen D, Cui QC, Yang H, Dou QP. Disulfiram, a clinically used anti-alcoholism drug and copper-binding agent, induces apoptotic cell death in breast cancer cultures and xenografts via inhibition of the proteasome activity. Cancer Res. 2006 Nov 1;66(21):10425-33. doi: 10.1158/0008-5472.CAN-06-2126. PMID 17079463
- [Background] Cvek B. Nonprofit drugs as the salvation of the world's healthcare systems: the case of Antabuse (disulfiram). Drug Discov Today. 2012 May;17(9-10):409-12. doi: 10.1016/j.drudis.2011.12.010. Epub 2011 Dec 16. PMID 22192884
- [Background] Suh JJ, Pettinati HM, Kampman KM, O'Brien CP. The status of disulfiram: a half of a century later. J Clin Psychopharmacol. 2006 Jun;26(3):290-302. doi: 10.1097/01.jcp.0000222512.25649.08. PMID 16702894
- See also: The trial status on sponsor's website. — http://imtm.cz/clinical-trials